CLINICAL TRIAL: NCT01976520
Title: NU 13H05: A Phase Ib Trial of Oncoquest-CLL Vaccine for Treatment-Naive Patients With Chronic Lymphocytic Leukemia
Brief Title: Vaccine Therapy for Treating Patients With Previously Untreated Chronic Lymphocytic Leukemia (CLL)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: XEME Biopharma Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 13H05; X12-11008 (Other: Theradex); P30CA060553 (NIH)
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: Cancer vaccine; Chronic lymphocytic leukemia; CLL; Autologous vaccine; B cell leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oncoquest-CLL vaccine treatment (Experimental): Patients receive Oncoquest-CLL vaccine subcutaneously on Day 1 and 15, and then monthly for 3 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Oncoquest-CLL vaccine

INTERVENTIONS:
Biological: Oncoquest-CLL vaccine — Comparison of 4 different dose levels of Oncoquest-CLL vaccine: 100 micrograms (mcg)/0.2 milliliters (mL), 200 mcg/0.4 mL, 375 mcg/0.75 mL, and 500 mcg/mL. Patients will receive a total of 5 doses of vaccines; the first 2 doses separated by 2 week intervals and the last 3 doses by 1 month intervals. Vaccine will be given by sc injections in 2 sites in upper arms or legs.
  Other Names: ATCE Vaccine, ATCEV, Autologous Tumor Vaccine, Oncoquest-CLL

SUMMARY:
This Phase I trial studies the safety and efficacy of vaccine therapy in treating patients with previously untreated chronic lymphocytic leukemia. Liposome-based vaccines containing an extract of a person's cancer cells and the immunostimulant interleukin-2 may help the body to build an effective immune response to kill cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of vaccination with Oncoquest-Chronic Lymphocytic Leukemia (CLL) vaccine (autologous tumor cell extract vaccine).

II. To evaluate the feasibility of Oncoquest-CLL production and administration to previously untreated patients with CLL.

SECONDARY OBJECTIVES:

I. To evaluate the clinical response [as defined by the International Workshop on Chronic Lymphocytic Leukemia 2008 (iwCLL2008)] of the Oncoquest-CLL vaccine in treatment-naive patients with CLL.

II. To evaluate the T and B cell immune responses against autologous leukemia cells induced with Oncoquest-CLL vaccine.

III. To measure the progression-free survival of patients treated with the Oncoquest-CLL vaccine.

IV. To evaluate the change in absolute lymphocyte count and lymphocyte doubling time before and after vaccine administration and correlate this with immune response.

OUTLINE:

Patients receive autologous tumor vaccine subcutaneously (SC) on Study Day 1 and 15, and then monthly for 3 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for 3 months, and then every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed B-CLL with low or intermediate risk disease as defined by the modified Rai criteria.
2. Patients must have lymphocytosis with white blood cells between 30,000-100,000/microliters (uL) in order to collect adequate leukemia cells for vaccine production.
3. Patients must have evidence of disease progression as demonstrated by an increase of more than 50% in lymphocytosis since diagnosis and/or lymphadenopathy and a lymphocyte doubling time of more than 6 months. Patients must have had at least 3 months of observation since diagnosis.
4. Patients must be age 18 years or older
5. Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Patients must have adequate renal and hepatic function:

   * Serum creatinine less than or equal to 2.0 mg/deciliter (dL)
   * Total Bilirubin less than or equal to 2.0 mg/dL
   * Serum glutamic-oxaloacetic transaminase/serum glutamate pyruvate transaminase (SGOT/SGPT) less than or equal to 2.5 x upper limit of normal (ULN)
7. Females of childbearing potential and sexually active males must consent to use of effective contraception. Child-bearing potential is defined as any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

   * Has not undergone a hysterectomy or bilateral oophorectomy; OR
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding consecutive 12 months).
8. All patients must have given signed, informed consent prior to registration on study.

Exclusion Criteria:

1. Patients who meet any of the NCI Working Group criteria to initiate treatment for CLL are NOT eligible for participation
2. Patients who have had or are currently receiving any treatment for CLL, including chemotherapy, corticosteroids, biologic therapy, or immunotherapy are NOT eligible for participation.
3. Patients who are actively receiving steroids or non-steroidal antiinflammatory drugs (NSAIDs) on a chronic basis and who are unwilling and/or unable to discontinue while on study therapy are NOT eligible for participation. NOTE: Patients must have discontinued steroids or NSAIDs for 1 week prior to registration to be considered eligible for participation.
4. Patients who are receiving cyclosporine, tacrolimus, or other chronic immunosuppressive agents are NOT eligible for participation.
5. Patients who exhibit any active or ongoing autoimmune processes including, but not limited to, autoimmune hemolytic anemia or immune thrombocytopenia purpura, are NOT eligible for participation.
6. Although rare, the only exception to this would be patients with Hashimoto's thyroiditis who ARE eligible for participation.
7. Patients who demonstrate the presence of antibodies to HIV or hepatitis C or presence of hepatitis B surface antigen or other active infectious process that could suppress the immune system and potentially interfere with the development of an immune response to the tumor antigen are NOT eligible for participation.
8. Patients who have a previous or concomitant malignancy are NOT eligible for participation EXCEPT for the following:

   * Patients with curatively treated squamous or basal cell carcinoma of the skin or effectively treated carcinoma in situ of the cervix ARE eligible for participation.
   * Patient who had a stage 1 solid tumor which has been adequately treated with curative intent, and has been in remission for more than 1 year.
   * Patients with a prior solid tumor who have been in remission more than 5 years ARE eligible for participation.
9. Patients who exhibit any significant concurrent, uncontrolled medical or psychiatric condition that in the opinion of the investigator would compromise the patient's ability to tolerate this treatment are NOT eligible for participation.
10. Patients who are pregnant or lactating are NOT eligible for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 30 days post-vaccination
  Safety data will be tabulated for all patients and include vital signs, laboratory parameters, and adverse events. Toxicities will be summarized descriptively by type and attribution.
Feasibility in terms of vaccine production. | Up to 4 weeks.
  The rate of successful production of the vaccine will be calculated. Successful production (feasibility) will be dichotomous. Dichotomous outcomes will be summarized using proportions and exact 95% binomial confidence intervals.
Feasibility in terms of vaccine delivery. | Up to 15 weeks.
  The rate of successful delivery of the vaccine will be calculated. Successful delivery (feasibility) will be dichotomous. Dichotomous outcomes will be summarized using proportions and exact 95% binomial confidence intervals.

SECONDARY OUTCOMES:
Clinical response evaluated using IWCLL2008 guidelines. | Up to 1 year.
  Clinical response to vaccination will be evaluated by parameters of reduction in leukemia cell count, lymph node size, liver and spleen size, and reduction in amount of disease in bone marrow) and improved hematologic parameters (including hemoglobin and platelet count).
In vitro immune response evaluated using T-cell and B-cell immune responses. | Up to 1 year.
  T-cell and B-cell responses will be summarized using medians and nonparametric confidence intervals.
Progression-free survival. | Up to 1 year.
Change in absolute lymphocyte count. | Baseline to up to 1 year.
Change in lymphocyte doubling time. | Baseline to up to 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Ma, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided